CLINICAL TRIAL: NCT06762600
Title: A Randomized, Double-Blind, Dose-Escalation, Placebo-Controlled Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Subcutaneous Injections of HRS-4729 Injection in Healthy Subjects
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of HRS-4729 Injection in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-4729-101
Record Dates: First submitted 2024-12-31; First posted 2025-01-07 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2024-12

CONDITIONS: Overweight or Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment group 1 (Experimental)
  Interventions: Drug: HRS-4729 injection; Drug: Acetaminophen
- Treatment group 2 (Placebo Comparator)
  Interventions: Drug: HRS-4729 injection placebo; Drug: Acetaminophen
- Treatment group 3 (Experimental)
  Interventions: Drug: HRS9531 injection
- Treatment group 4 (Placebo Comparator)
  Interventions: Drug: HRS9531 injection placebo

INTERVENTIONS:
Drug: HRS-4729 injection — HRS-4729 injection
  Arms: Treatment group 1
Drug: HRS-4729 injection placebo — HRS-4729 injection placebo
  Arms: Treatment group 2
Drug: HRS9531 injection — HRS9531 injection
  Arms: Treatment group 3
Drug: HRS9531 injection placebo — HRS9531 injection placebo
  Arms: Treatment group 4
Drug: Acetaminophen — Acetaminophen
  Arms: Treatment group 1; Treatment group 2

SUMMARY:
The study is being conducted to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of HRS-4729 injection in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily provides written informed consent prior to the initiation of any study-related activities and demonstrates understanding of the procedures and methods involved in the study, agreeing to adhere strictly to the clinical trial protocol to complete the study.
2. Male or female subjects; aged 18 to 55 years.
3. Self-reports no more than a 5 kg change in body weight during the 3 months prior to screening (including the screening visit).

Exclusion Criteria:

1. A history of current significant disease in the neurological, psychiatric, cardiovascular, gastrointestinal, respiratory, genitourinary, endocrine, hematologic, or immune systems, as determined by the investigator, which would render the subject unsuitable for participation in this trial.
2. A history of significant gastrointestinal disease or related symptoms, conditions affecting gastric emptying, or prior gastrointestinal surgery.
3. Subjects who have had a major surgery or severe trauma within 6 months prior to screening, or who are planned for surgical procedures during the trial period.
4. Participation in any drug or medical device clinical trial within 3 months prior to screening.
5. Any abnormal physical examination, vital signs, laboratory tests, chest X-ray and abdominal ultrasound findings deemed clinically significant by the investigator, rendering the subject unsuitable for participation.
6. Clinically significant abnormalities on 12-lead ECG as determined by the investigator.
7. Known or suspected history of drug abuse or substance dependence, or positive urine drug screen during the screening period.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 103 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | Screening period up to day 43.

SECONDARY OUTCOMES:
The maximum plasma concentration (Cmax) | Post-dose at day 1 to day 43.
Time to maximum plasma concentration (Tmax) | Post-dose at day 1 to day 43.
Terminal half-life (t1/2) | Post-dose at day 1 to day 43.
Apparent clearance (CL/F) | Post-dose at day 1 to day 43.
Apparent volume of distribution (Vz/F) | Post-dose at day 1 to day 43.
Anti-HRS-4729 antibodies | Post-dose at day 1 to day 43.
Changes from baseline in Fasting Body Weight | Run-in Period up to Day 113.
Changes from baseline in Fasting Plasma Glucose | Run-in Period up to Day 113.
Changes from baseline in Fasting Insulin | Run-in Period up to Day 113.
Changes from baseline in Fasting C-Peptide | Run-in Period up to Day 113.
Total fat mass | Run-in Period up to Day 113.

CONTACTS AND LOCATIONS:
Locations (1):
- Jinan Central Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided